CLINICAL TRIAL: NCT01231269
Title: Whole-body Diffusion-weighted Magnetic Resonance Imaging for Staging and Treatment Prediction of Lymphoma
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: S51160
Record Dates: First submitted 2010-10-28; First posted 2010-11-01 (Estimated); Last update posted 2024-07-10 (Actual); Status verified 2024-07

CONDITIONS: Lymphoma; Hodgkin Lymphoma; Non-Hodgkin Lymphoma (Follicular, Diffuse B-cel Lymphoma, PTLD and Mantle Cel Lymphoma)
MeSH Terms: conditions — Lymphoma; Hodgkin Disease; Lymphoma, Non-Hodgkin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- MRI (Experimental): diffusion-weighted MRI
  Interventions: Other: MRI

INTERVENTIONS:
Other: MRI — MRI scan without administration of contrast/without radiation

SUMMARY:
Whole body diffusion-weighted imaging is a functional magnetic resonance imaging technique that characterizes tissue by probing changes in water diffusion secondary to differences in the tissue microstructure. These changes in water diffusion result in differences in signal intensity on diffusion-weighted-images that are quantified with the apparent diffusion coefficient (ADC). In malignant lesions, the extravascular extracellular space (EES) will be diminished, due to the increased number of cells. This will restrict water diffusion, identified by increased signal intensity (SI) on native DWI images and low ADC. Several studies indicate the value of DWI for differentiation of benign and malignant lymph nodes, detection of tumor recurrence and for ADC-based prediction of treatment outcome in various solid tumours (Koh DM et al, Am J Roentgenol 2007).

Patients with a new diagnosis of Hodgkin or Non-Hodgkin Lymphoma (only diffuse large B-cell lymphoma, follicular lymphoma, mantle cell lymphoma and PTLD) will be included in the study. These patients will receive a WB-DWI scan before treatment, once or twice during treatment (depending on the type of lymphoma) and after the completion of the treatment. The MRI scan will be performed on a 3 Tesla-MRI system without contrast administration and without exposing the patient to radiation.

Whole body diffusion-weighted images will be prospectively interpreted by two experienced radiologists, blinded to all clinical and imaging data. Findings will be correlated to FDG-18F-2-fluoro-2-deoxy-D-glucose fluorodeoxyglucose , biopsies performed in clinical routine (bone marrow always - soft tissue lesions if indicated) and imaging follow-up.

The purpose of this study is:

* to evaluate Whole body diffusion-weighted imaging for staging of lymphoma
* to evaluate Whole body diffusion-weighted imaging as an early predictive biomarker for treatment outcome
* to evaluate Whole body diffusion-weighted imaging for differentiating residual tumor from post therapy changes

ELIGIBILITY:
Inclusion Criteria:

* every patient with a new diagnosis of Hodgkin or Non-Hodgkin Lymphoma (only diffuse large B-cel lymphoma, mantle cell lymphoma, follicular lymphoma and PTLD)

Exclusion Criteria:

* patient with general contraindications for MRI (pacemaker, claustrophobia, etc.)
* patients with a type of lymphoma other than those described in the inclusion criteria

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2010-11 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
disease stage | 4 years
  Lesions are characterized as benign or malignant based on signal intensity and ADC values, enabling correct determination of tumor extent (staging).

SECONDARY OUTCOMES:
progression free survival | 6 years
  We will investigate whether there is a correlation between ADC and signal intensity changes during therapy and progression free survival

CONTACTS AND LOCATIONS:
Overall Officials: vincent vandecaveye, MD PhD, Principal Investigator — Universitaire Ziekenhuizen KU Leuven
Locations (1):
- University Hospital Leuven, Leuven, Vlaams-Brabant, Belgium

REFERENCES:
- [Derived] De Paepe KN, Van Keerberghen CA, Agazzi GM, De Keyzer F, Gheysens O, Bechter O, Wolter P, Dierickx D, Janssens A, Verhoef G, Oyen R, Koole M, Vandecaveye V. Quantitative Whole-Body Diffusion-weighted MRI after One Treatment Cycle for Aggressive Non-Hodgkin Lymphoma Is an Independent Prognostic Factor of Outcome. Radiol Imaging Cancer. 2021 Mar 26;3(2):e200061. doi: 10.1148/rycan.2021200061. eCollection 2021 Mar. PMID 33817648